CLINICAL TRIAL: NCT06850987
Title: Evaluation of the Effects of Nonsurgical Periodontal Treatment on Apelin and Oxidative Stress Levels in Individuals With Periodontitis
Brief Title: Effect of Nonsurgical Periodontal Treatment on Apelin and Oxidative Stress Levels
Status: Completed | Type: Observational
Sponsor: Hatice Yemenoğlu (Other)
Collaborators: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Sponsor-Investigator, Hatice Yemenoğlu, Principal investigator, Recep Tayyip Erdogan University Training and Research Hospital
Organization: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Other Study IDs: Recep TayyipErdoganUniversity
Record Dates: First submitted 2025-02-16; First posted 2025-02-28 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Stage 1-2 periodontitis group
  Interventions: Procedure: non surgical periodontal therapy; Other: measurement of periodontal clinical parameters; Other: Gingival crevicular fluid samples will be collected
- Stage 3-4 periodontitis group
  Interventions: Procedure: non surgical periodontal therapy; Other: measurement of periodontal clinical parameters; Other: Gingival crevicular fluid samples will be collected

INTERVENTIONS:
Procedure: non surgical periodontal therapy — All participants will have their non-surgical periodontal treatments completed after samples are taken and periodontal measurements are taken at the beginning.
Other: measurement of periodontal clinical parameters — Periodontal measurements will be taken from all participants at baseline, 1 month, 3 months and 6 months
Other: Gingival crevicular fluid samples will be collected — Gingival crevicular fluid samples will be collected from all participants at baseline, 1 month, 3 months and 6 months

SUMMARY:
Periodontitis is a multifactorial, chronic inflammatory disease triggered by microorganisms in the dental biofilm. The limited data of clinical periodontal measurements in the diagnosis of periodontitis have led to the search for more reliable biomarkers that can be used in the diagnosis and follow-up of periodontal diseases. Apelin is another adipokine that has been investigated in a small number of studies so far; its receptor (apelin reseptor (APJ)) was first identified in 1993 and later isolated as a molecule in 1998. Studies have focused on this form of apelin-13 due to its high biological activity. Although apelin-13 is considered the most biologically active form, it has been shown that apelin-36 has a much higher binding affinity to APJ than apelin-13. Periodontitis is the most common cause of tooth loss in adults, and is associated with systemic conditions such as metabolic syndrome, diabetes mellitus, and cardiovascular disease. The elucidation of these possible interactions has been the focus of many studies. Apelin is associated with insulin secretion, as well as its effects on lipid and glucose metabolism. Studies in both humans and animals have shown that type 2 diabetes and obesity are typically associated with increased plasma apelin levels. Based on this observation, recent studies have shown that salivary and serum apelin levels are higher in individuals with chronic periodontitis and type 2 diabetes compared to healthy individuals. Considering all this information, the investigators considered that apelin may be a biomarker for periodontal diseases due to its inflammation-regulating effects as a result of the change in gingival crevicular fluid (GCF) apelin-13, apelin-36 and total oxidant status (TOS)/total antioxidant status (TAS) levels compared to the initial level after non-surgical periodontal treatment in systemically healthy and periodontitis individuals, considering the relationship of adipokines with periodontal disease in this study.

ELIGIBILITY:
Inclusion Criteria:

* Being systemically healthy
* Not smoking
* Not using anti-inflammatory drugs in the last 3 months, antibiotics and systemic corticosteroids in the last 6 months
* Not being pregnant or lactating
* Not having received periodontal treatment in the last 6 months
* Having at least 20 teeth in the mouth
* Being diagnosed with periodontitis (Stage 1-2 and Stage 3-4) by the researcher

Working groups will be formed based on the 2017 Periodontal Disease Classification

Exclusion Criteria:

being periodontally healthy having systemic disease being pregnant and lactating smoking having periodontal treatment in the last 6 months having fewer than 20 teeth

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: periodontitis
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-08-16 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2025-06-14 (Actual)

PRIMARY OUTCOMES:
Periodontal pocket depth | at baseline, 1 month, 3 months and 6 months
  It will be calculated by measuring the distance between the gingival margin and the pocket base. Each tooth will be measured from six surfaces and averaged. higher scores indicate worse outcome.
clinical attachment loss | at baseline, 1 month, 3 months and 6 months
  It will be calculated by measuring the distance between the cementoenamel border and the pocket base. It will be measured from the six surfaces of each tooth and the average will be taken. higher scores indicate worse outcome.

SECONDARY OUTCOMES:
Apelin-13 level | at the beginning, at 1 month, at 3 months and at 6 months
  Determination of the levels of apelin-13 from gingival crevicular fluid (GCF) samples will be done by ELISA method
Apelin-36 level | at baseline, 1 month, 3 months and 6 months
  Determination of the levels of apelin-36 from gingival crevicular fluid (GCF) samples will be done by ELISA method
TOS (total oxidant status) level | at baseline, 1 month, 3 months and 6 months
  Determination of the levels of TOS (total oxidant status) from gingival crevicular fluid (GCF) samples will be done by ELISA method
TAS (total antioxidant status) level | at baseline, 1 month, 3 months and 6 months
  Determination of the levels of TAS (total antioxidant status) from gingival crevicular fluid (GCF) samples will be done by ELISA method

CONTACTS AND LOCATIONS:
Locations (1):
- Recep Tayyip Erdoğan University Faculty of Dentistry, Rize, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
If deemed necessary, necessary information can be provided to protect patient confidentiality.
Supporting Information: Study Protocol, SAP